CLINICAL TRIAL: NCT06971029
Title: Effects Of Supplementation With New Technology for Obtaining Low Molecular Weight Hydrolyzed Collagen Vs. Verisol Collagen on Expression Lines, Skin Quality in the Orbicularis Oculi Region, And Serum Levels of Klotho, VEGF, and TGF-Beta
Brief Title: IMPACT OF SUPPLEMENTATION WITH LOW MOLECULAR WEIGHT HYDROLYZED COLLAGEN AND VERISOL ON THE EXPRESSION OF LINES, SKIN QUALITY, AND LEVELS OF KLOTHO, VEGF, AND TGF-BETA IN THE EYE REGION
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodolfo de Paula Vieira, Prof. Dr., Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7.233.377
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Skin Health; Collagen Supplementation; Growth Factors
Keywords: Skin health; collagen supplementation; growth factors
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: The 150 volunteers will be randomized into three groups (n = 50/group): Verisol Collagen 2.5 g/day (GCV), Peptech Collagen 2.5 g/day (GCP 2.5), and Peptech Collagen 10 g/day (GCP 10).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Verisol Collagen 2.5 g/day (Experimental): Supplementation with Verisol® collagen will be administered at a dose of 2.5 g/day, diluted in water or water-based juice (300-500 mL), and should be consumed daily, 7 days a week, for 3 months.
  Interventions: Dietary Supplement: Supplementation with Verisol®
- Peptech Collagen 2.5 g/day (GCP 2.5) (Experimental): Supplementation with Peptech® collagen will be administered at a dose of 2.5 g/day, diluted in water or water-based juice (300-500 mL), and should be consumed daily, 7 days a week, for 3 months.
  Interventions: Dietary Supplement: Supplementation with Peptech® 2.5G
- eptech Collagen 10 g/day (GCP 10) (Experimental): Supplementation with Peptech® collagen will be administered at a dose of 10.0 g/day, diluted in water or water-based juice (300-500 mL), and should be consumed daily, 7 days a week, for 3 months.
  Interventions: Dietary Supplement: Supplementation with Peptech® 10.0G
- Group Control (Other): he control group will undergo the tests but will not receive supplementation.
  Interventions: Diagnostic Test: Control group

INTERVENTIONS:
Dietary Supplement: Supplementation with Verisol® — Supplementation with Verisol® collagen will be administered at a dose of 2.5 g/day, diluted in water or water-based juice (300-500 mL), and should be consumed daily, 7 days a week, for 3 months.
  Arms: Verisol Collagen 2.5 g/day
Dietary Supplement: Supplementation with Peptech® 2.5G — Supplementation with Peptech® collagen will be administered at a dose of 2.5 g/day, diluted in water or water-based juice (300-500 mL), and should be consumed daily, 7 days a week, for 3 months.
  Arms: Peptech Collagen 2.5 g/day (GCP 2.5)
Dietary Supplement: Supplementation with Peptech® 10.0G — Supplementation with Peptech® collagen will be administered at a dose of 10.0 g/day, diluted in water or water-based juice (300-500 mL), and should be consumed daily, 7 days a week, for 3 months.
  Arms: eptech Collagen 10 g/day (GCP 10)
Diagnostic Test: Control group — The control group will not receive supplementation.
  Arms: Group Control

SUMMARY:
Skin is the largest organ of the human body and performs various vital functions, including protection against external agents, regulation of body temperature, and sensory perception. As we age, our skin undergoes a series of changes that can be noticeable both visually and physically. One of the most evident changes is the appearance of wrinkles and fine lines, resulting from decreased skin elasticity and reduced production of collagen and elastin. Nutrition plays a key role in skin health, influencing its structure, function, and ability to defend against damage and diseases. However, it is unknown to what extent supplementation with different types of collagens can attenuate these effects in middle-aged women. Therefore, the present study aims to recruit 150 middle-aged women (35-58 years old) who will be randomized into three groups, Verisol Collagen 2.5 g/day, Peptech Collagen 2.5 g/day, and Peptech Collagen 10 g/day, 7 days a week, for 3 months. Skin hydration, oiliness, and flexibility, as well as the number and depth of expression lines, will be evaluated, along with plasma levels of Klotho, VEGF, and TGF-beta. Data will be analyzed, and graphs constructed using GraphPad Prism 5.0 software (California, USA). The normality distribution of the data will be assessed by the Kolmogorov-Smirnov test. Data with parametric distribution will be subjected to paired Student's t-test for intragroup comparison, and unpaired t-test will be used for comparison between groups. Significance levels will be considered statistically different for p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* "Inclusion criteria require that volunteers be between 35 and 58 years old, have been sedentary for at least one year, and, after reading and understanding all stages of the study, agree to and sign the informed consent form (ICF).

Exclusion Criteria:

* "Exclusion criteria include undergoing facial aesthetic procedures involving hyaluronic acid or botulinum toxin, being an active or passive smoker within the past 3 years, using protein- or amino acid-based supplements within the past 6 months, or using cosmetics with skin-repairing properties in the orbicularis oculi region.

Ages: 35 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2025-06-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of Klotho, VEGF, and TGF-beta | Three months.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Proksch E, Brandner JM, Jensen JM. The skin: an indispensable barrier. Exp Dermatol. 2008 Dec;17(12):1063-72. doi: 10.1111/j.1600-0625.2008.00786.x. PMID 19043850
- [Derived] Paula-Vieira RHR, Dias SR, Silva-Reis A, Moura-Maia MS, Ramos-Gomes NV, Jesus-Silva K, Oliveira-Leal YR, Castro-Pimentel LT, Carvalho WSF, Melo F, Martins JLR, Bachi ALL, Vieira RP. Immune-Modulatory Effects of Bioactive Collagen Peptides Improve Skin Health in Middle-Aged Women. Dermatol Ther (Heidelb). 2026 Jan 27. doi: 10.1007/s13555-026-01654-9. Online ahead of print. PMID 41588262